CLINICAL TRIAL: NCT05430958
Title: Phase 1 Open Label Study to Evaluate the Safety, Tolerability, and Immunogenicity of an Intradermal Booster Dose of INO-4800 Alone or in Combination With INO-9112 Followed by Electroporation, in Adults Who Completed a Primary Immunization Series Against SARS-CoV-2 With mRNA Vaccines
Brief Title: Safety, Tolerability and Immunogenicity of INO-4800 for COVID19 in Healthy Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was withdrawn due to sponsor decision.
Sponsor: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COVID19-131
Record Dates: First submitted 2022-06-21; First posted 2022-06-24 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Coronavirus Infection
Keywords: DNA vaccine; Coronavirus Infection; SARS-CoV-2; COVID19
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — reluscovtogene ralaplasmid; rocakinogene sifuplasmid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (8):
- Group 1 (Experimental): Single injection of 0.8 mg of INO-4800 followed by EP administered at Day 0
  Interventions: Drug: INO-4800; Device: CELLECTRA® 2000
- Group 2 (Experimental): Single injection of 0.8 mg of INO-4800 plus 0.05 mg of INO-9112 followed by EP administered at Day 0
  Interventions: Drug: INO-4800; Drug: INO-9112; Device: CELLECTRA® 2000
- Group 3 (Experimental): Single injection of 0.8 mg of INO-4800 plus 0.10 mg of INO-9112 followed by EP administered at Day 0
  Interventions: Drug: INO-4800; Drug: INO-9112; Device: CELLECTRA® 2000
- Group 4 (Experimental): Single injection of 0.8 mg of INO-4800 plus 0.20 mg of INO-9112 followed by EP administered at Day 0
  Interventions: Drug: INO-4800; Drug: INO-9112; Device: CELLECTRA® 2000
- Group 5 (Experimental): Two injections of 0.8 mg (1.6 mg total) of INO-4800 followed by EP administered at Day 0
  Interventions: Drug: INO-4800; Device: CELLECTRA® 2000
- Group 6 (Experimental): Two injections of 0.8 mg (1.6 mg total) of INO-4800 + 0.05 mg (0.1 mg total) of INO-9112 followed by EP administered at Day 0
  Interventions: Drug: INO-4800; Drug: INO-9112; Device: CELLECTRA® 2000
- Group 7 (Experimental): Two injections of 0.8 mg (1.6 mg total) of INO-4800 + 0.1 mg (0.20 mg total) of INO-9112 followed by EP administered at Day 0
  Interventions: Drug: INO-4800; Drug: INO-9112; Device: CELLECTRA® 2000
- Group 8 (Experimental): Two injections of 0.8 mg (1.6 mg total) of INO-4800 + 0.20 mg (0.40 mg total) of INO-9112 followed by EP administered at Day 0
  Interventions: Drug: INO-4800; Drug: INO-9112; Device: CELLECTRA® 2000

INTERVENTIONS:
Drug: INO-4800 — INO-4800 will be given at 0.8 or 1.6 mg for at least 6 months but no more than 12 months following the completion of a primary vaccination.
Drug: INO-9112 — INO-9112 will be given in at various doses (dose of 0, 0.05, 0.10, 0.20 or 0.40 mg) in combination with INO-4800.
  Arms: Group 2; Group 3; Group 4; Group 6; Group 7; Group 8
Device: CELLECTRA® 2000 — Electroporation (EP) using the CELLECTRA® 2000 device will be administered following ID delivery of INO-4800.

SUMMARY:
This is an open label, phase 1 clinical trial of an intra-dermal booster dose of INO-4800 alone or in combination with INO-9112 followed by electroporation (EP) among healthy adults at least 18 years of age, who previously completed their primary immunization series with mRNA vaccines against SARS-CoV-2 within 6-12 months prior to the booster dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and non-pregnant women at least 18 years of age;
* Able and willing to comply with all study procedures;
* Screening laboratory results within normal limits or deemed not clinically significant by the Investigator;
* Received full primary series doses of an approved or authorized mRNA vaccine at least 6 months but no more than 12 months prior to INO-4800 booster dose.
* Must meet one of the following criteria with respect to reproductive capacity:

  * Women who are post-menopausal as defined by reported spontaneous amenorrhea for ≥ 12 months;
  * Surgically sterile (i.e., vasectomy in males or tubal ligation, absence of ovaries and/or uterus in females). In the case of vasectomy, participants should wait six (6) months post-vasectomy prior to enrollment;
  * Use of medically effective contraception with a failure rate of < 1% per year when used consistently and correctly from screening until Day 28 post booster dose.

Exclusion Criteria:

* Acute febrile illness with temperature >100.4°F (38.0°C) or acute onset of upper or lower respiratory tract symptoms (e.g., cough, shortness of breath, sore throat) within the prior 72 hours;
* Positive SARs-CoV-2 PCR test, if results are available prior to dosing;
* Pregnant or breastfeeding, or intending to become pregnant or intending to father children within the projected duration of the study starting from the Screening visit until Day 28 post booster dose;
* Positive pregnancy test during screening or immediately prior to booster dose;
* Positive HIV rapid test, Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody at Screening;
* Is currently participating or has participated in a study with an IP within 30 days preceding Day 0 (documented receipt of placebo in a previous study would be permissible for study eligibility);
* Currently participating in another study with an investigational product during the conduct of this study;
* Previous or planned receipt of any COVID-19 booster vaccine during the trial period
* Medical conditions as follows:

  * Respiratory diseases
  * History of hypersensitivity or severe allergic reaction
  * Uncontrolled hypertension
  * Uncontrolled diabetes mellitus
  * Malignancy within the past 2 years, with the exception of superficial skin
  * History of cardiovascular disease
  * History of myocarditis or pericarditis
  * History of seizures within the past 2 years
  * Underlying immunosuppressive illness
* Lack of acceptable sites for ID injection and EP
* Blood donation or transfusion within 1 month prior to Day 0;
* Reported alcohol or substance abuse/dependence or illicit drug use within the past year;
* Any non-study vaccine (e.g., influenza vaccine) within 2 weeks prior to the dose of IP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Solicited Local and Systemic Adverse Events (AEs) | Baseline up to Day 7
Percentage of Participants with Adverse Events (AEs) | Baseline up to Day 28
Percentage of Participants with Serious Adverse Events (SAEs) | Baseline up to week 52
Percentage of Participants with Adverse Events of Special Interest (AESIs) | Baseline up to week 52
Percentage of Participants with Incidence of medically attended AEs (MAAEs) | Baseline up to week 52
Percentage of Participants with Change in SARS-CoV-2 pseudovirus neutralizing titers | Baseline up to day 28

SECONDARY OUTCOMES:
Number of Participants with a Change in SARS-CoV-2 pseudovirus neutralizing titers | Baseline, Day 7, 14, 84, 180, 224, 280 and 365 post-booster
Number of Participants with SARS-CoV-2 pseudovirus neutralizing titers | Days 7, 14, 28, 84, 180, 224, 280 and 365 post-booster
Number of Participants with ARS-CoV-2 Spike binding IgG and change in SARS-CoV-2 Spike binding IgG | Days 7, 14, 28, 84, 180 and 365 post-booster
Number of Participants with SARS-CoV-2 cellular immune response as measured by IFN-gamma ELISpot | Day 14 post-booster

CONTACTS AND LOCATIONS:
Overall Officials: Jose Suaya, MD, Study Director — Inovio Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No